CLINICAL TRIAL: NCT00459329
Title: PEARL Intervention to Reduce Depression Among Adults With Epilepsy
Acronym: PEARL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Paul Ciechanowski, MD, MPH, University of Washington
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 06-4237-C 01; NCT00459329; SIP 07-2006
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Depression; Epilepsy
Keywords: Depression; Epilepsy; Problem-Solving Therapy; Mental Health; Neurology; Home-based health care; Community-based program; Collaborative care
MeSH Terms: conditions — Depression; Epilepsy; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Program to Encourage Active, Rewarding Lives (PEARL) — Eight 50-minute in-home sessions over 19 weeks with a masters-level social work counselor using Problem Solving Therapy (PST).
  PST is a skills-enhancing behavioral depression treatment based on the assumption that an accumulation of problems in living cause and maintain depressive symptoms, and through systematically identifying and addressing these problems, patients achieve decreased depressive symptoms. Counselors also help participants to increase social and physical activities and to incorporate pleasant activities into patients' lives.
  Counselors provide education and monitoring for antidepressant use, and work with the participant's physician and PEARL psychiatrist to recommend initiating or adjusting antidepressant medications. The PHQ-9 is administered at each session to track depression change.
  After 19 weeks, counselors will maintain monthly telephone calls with participants, administering the PHQ-9 and assessing PST success.

SUMMARY:
The purpose of this study is to test the effectiveness of a home-based depression treatment intervention called "Program to Encourage Active, Rewarding Lives (PEARL)". We hypothesize that over a 12-month period, compared to usual care, those receiving the PEARL intervention will show more improvement with their depression, have higher quality of life and function, and use fewer medical services.

DETAILED DESCRIPTION:
Compared to non-depressed individuals with epilepsy, those with depression have significantly higher rates of suicide, lower social and occupational functioning, decreased quality of life independent of seizure frequency, and higher non-psychiatric health care utilization. Adults with epilepsy are more likely to be homebound as a result of reduced function and restrictions in driving, opportunities to obtain enhanced quality of care for depression may be limited. This study tests the effectiveness of a home-based multi-modal depression treatment intervention called Program to Encourage Active, Rewarding Lives (PEARL). PEARL consists of problem solving treatment, social and physical activation, pleasant events scheduling, support and education regarding antidepressant medication use as well as psychiatric consultation and recommendations regarding initiation or adjustment of antidepressant medications.

In a sample of adults with epilepsy who have minor depression, major depression and/or dysthymia, we hypothesize that over a 12-month period, compared to usual care, those randomized to the PEARL intervention will: achieve higher levels of depression response and remission, achieve higher quality of life and function, and utilize less non-psychiatric health care.

By providing a multi-modal, home-based stepped collaborative care intervention for adults with depression and epilepsy, this program will offer practical alternatives to usual care and will provide a program for improving depression outcomes, quality of life and potentially, epilepsy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Home address within 30 miles of Seattle
* Diagnosis of epilepsy (ICD-9 code 345.XX)
* Appointment in the UW REC or Neurology clinic in the past 2 years and currently enrolled in this clinic.
* Current age older than 18 years
* Diagnosis of major depression, minor depression or dysthymia
* Ability to speak/read English

Exclusion Criteria:

* Alcohol and/or substance abuse/dependence based on a score greater than 1 on 4-item validated CAGE-AID
* Cognitive impairment based on a score less than 3 on a 6-item validated cognitive screen
* Diagnosis of bipolar disorder, schizophrenia/schizoaffective disorder or other psychotic disorder
* Women who are pregnant or nursing
* Terminal medical illness
* Those currently seeing or planning to see a psychiatrist
* Those with suicidal ideation nearly every day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Mean SCL-20 depression scores | 6 & 12 months post-baseline
Depression treatment response, defined as greater than 50% decrease in SCL-20 score from baseline | 6 & 12 months post-baseline
Complete depression remission defined as SCL-20 score less than 0.5. | 6 & 12 months post-baseline

SECONDARY OUTCOMES:
Quality of Life | 6 & 12 months post-baseline
Pharmaceutical and health care utilization and costs | 6 & 12 months post-baseline
Seizure frequency and severity | 6 & 12 months post-baseline
Satisfaction with epilepsy health care | 6 & 12 months post-baseline
Epilepsy Self-Efficacy | 6 & 12 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Ciechanowski, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Regional Epilepsy Center, Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Chaytor N, Ciechanowski P, Miller JW, Fraser R, Russo J, Unutzer J, Gilliam F. Long-term outcomes from the PEARLS randomized trial for the treatment of depression in patients with epilepsy. Epilepsy Behav. 2011 Mar;20(3):545-9. doi: 10.1016/j.yebeh.2011.01.017. Epub 2011 Feb 18. PMID 21333607
- [Derived] Ciechanowski P, Chaytor N, Miller J, Fraser R, Russo J, Unutzer J, Gilliam F. PEARLS depression treatment for individuals with epilepsy: a randomized controlled trial. Epilepsy Behav. 2010 Nov;19(3):225-31. doi: 10.1016/j.yebeh.2010.06.003. Epub 2010 Jul 6. PMID 20609631